CLINICAL TRIAL: NCT06587854
Title: a PRagmatic Observational Study of Congestion proFILes in patiEnts With Acute Heart
Brief Title: a PRagmatic Observational Study of Congestion proFILes in patiEnts With Acute Heart Failure
Acronym: PROFILE-AHF
Status: Recruiting | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Jozine ter Maaten, Principal Investigator, University Medical Center Groningen
Other Study IDs: 20486
Record Dates: First submitted 2024-08-25; First posted 2024-09-19 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Acute Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood: blood samples from different time points will be collected and stored, for later further analysis Urine: urine samples will be collected and stored, for later further analysis
  As part of substudy:
  Skin biopsy: A skin biopsy is collected, with one portion processed for analysis of sodium and water storage, while another portion is used to determine glycosaminoglycan levels
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational is to study the prevalence of distinct congestion phenotypes and study their association with response to therapy and outcomes in acute heart failure patients. The main question[s] it aims to answer [is/are]:

* Primary objective: to study the prevalence of distinct congestion phenotypes
* Other objectives (including):

  * Response to therapy as assessed by

    * Natriuresis after 24 hours
    * Rehospitalization and/or deats after 6 months
  * Length of hospital stay
  * Congestion at discharge
  * Changes in filling pressures over time
  * Relationship between liver stiffness, as assessed with Fibroscan and congestion
  * Substudy: glycosaminoglycan netword and endothial glycocalyx

Participants will undergo several extra study related measurements:

* Assessment of filling pressures with ultrasound
* Ultrasound investigation of the lungs and kidneys
* Fibroscan of the liver
* Sidestream darkfield imaging sublingual
* As part of substudy GLYCO-AHF: skin biopsy to determine glycocalyx, as well as salt and water content.
* As part of substudy PREACH-AHF: the effects of peripheral venous congestion and endothelial dysfunction on a large screen of plasma proteins

DETAILED DESCRIPTION:
Objective: to study the prevalence of distinct congestion phenotypes and investigate their association with response to therapy and outcomes in acute heart failure patients.

Study design: Observational, prospective study

Study population: 270 patients admitted with the primary diagnosis of acute heart failure requiring intravenous loop diuretics.

Main study parameters/endpoints:

To identify distinct congestion phenotypes and study their association with response to therapy and outcomes

Secondary outcomes: total natriuresis after 24 hours, and first occurrence of all-cause mortality or heart failure rehospitalisation at 6 months Exploratory outcomes include: length of hospital stay, congestion at discharge and changes in filling pressures over time. Furthermore, as part of the GLYCO-AHF substudy: the expression of glycosaminoglycans and, as part of the PREACH-AHF substudy: the effects of peripheral venous congestion and endothelial dysfunction on a large screen of plasma proteins.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to give written informed consent
* Age ≥ 18 years
* Male or female
* Primary diagnosis of acute heart failure at presentation, with signs and symptoms of tissue decongestion. Diagnosis is based on the criteria in the ESC HF guidelines (1)
* Requirement of intravenous loop diuretics

Exclusion Criteria:

* Patients with severe kidney dysfunction (in need for ultrafiltration or dialysis)
* Previous participation in this study
* Inability to follow instructions
* Dyspnoea or oedema primarily due to non-cardiac causes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients admitted to the hospital with a primary diagnosis of acute heart failure
Sampling Method: Probability Sample
Enrollment: 270 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
To study the prevalence of distinct congestion phenotypes | From date of hospital admission untill the date of discharge (from this admission), with an expected discharge after 5 to 10 days after admission.
  Based on the degree of congestion and edema in combination with intravascular pressures, patients will be classified into different phenotypes (high/low intravascular pressures and extensive/minimal edema.

SECONDARY OUTCOMES:
Total natriuresis after 24 hours | 24 hours
  To assess this, urine is collected for 24 hours after the first administration of diuretics according to the hospital protocol and natriuresis is calculated as the total amount of diuresis (L) multiplied by the urinary sodium concentration (mmol/L).with natriuresis as the primary outcome measure.
Rehospitalization and/or death after 6 months | 180 days

OTHER OUTCOMES:
Congestion at discharge | Date of discharge, or maximum two days before. Expected to be between 5-10 days after admission.
  Congestion at discharge will be assessed by several measures; clinical symptoms (e.g. orthopnoea, dyspnoea), physical examination (e.g. oedema, rales, jugular venous pressure), ultrasound examination (lungs, heart, inferior vena cava,.
Changes in filling pressures over time | From date of hospital admission untill the date of discharge, or maximum two days before. Expected to be between 5-10 days after admission.
  Using either a Swan Ganz catheter (if present as part of standard of care) or echocardiography, intravasculair filling pressures will be measured daily.
Length of stay | Variable, from date of admission untill date of discharge. Expected to be between 5-10 days after admission.
  Number of days of the index hospitalization
Liver stiffness, as assessed with Fibroscan | From date of hospital admission untill the date of discharge, or maximum two days before. Expected to be between 5-10 days after admission.
  Congestion of the liver reflected by liver stifness will be determined after admission and at discharge (with maximum two days before).
Differences in microvasculature | From date of hospital admission untill the date of discharge, or maximum two days before. Expected to be between 5-10 days after admission.
  Subligual sidestream darkfield imaging will be performed at day 1 or 2 and will be repeated at discharge (or maximum two days before). This technique allows for a detailed observation of capillary blood flow, capillary density and glycocalyx integrity. Comparing the microvasculature between the different congestion phenotype groups, as well as studying changes in the microvasculature from admission to discharge will provide novel information with regards to the microvasculature in AHF patients.
(Substudy GLYCO-AHF): Differences in glycosaminoglycan network | From date of hospital admission untill the date of discharge, or maximum two days before. Expected to be between 5-10 days after admission.
  A skin biopsy will be performed at day 1 or 2. At discharge, or maximum two days before, patients will receive a second skin biopsy. With the biopsy the glycosaminoglycan network and glygocalyx can be determined. Cryosections will be stained using available antibodies for glycosaminoclycans, whereafter their immunochemical expression will be quantified. The expression will be compared between both the different patient groups (based on phenotype) as well as between the two biopsies (at admission and at discharge).
(Substudy PREACH-AHF): Effects of peripheral venous congestion on plasma proteins | Date of discharge, or maximum two days before.
  To study the effect of peripheral venous congestion and endothelial dysfunction on plasma proteins, blood samples will be taken via an intravenous line before and after inflating a pressure cuff, while a pressure transducer measures the peripheral venous pressure. Patients will also undergo a reactive hyperaemia index measurement to investigate the link between plasma proteins and endothelial dysfunction. These measurements will be performed at discharge or a maximum of 2 days before.

CONTACTS AND LOCATIONS:
Locations (1):
- UMCG, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No